CLINICAL TRIAL: NCT06791304
Title: Effectiveness of Doppler Renal Resistive Index in Early Detection of Postoperative Acute Kidney Injury in Prolonged Cardiopulmonary Bypass Cardiac Surgeries
Brief Title: Renal Resistive Index in Early Detection of Postoperative Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Musa Harun UÇAR, anesthesiology and reanimation doctor, Bursa Yuksek Ihtisas Training and Research Hospital
Other Study IDs: 2011-KAEK-25 2022/08-16
Record Dates: First submitted 2024-12-27; First posted 2025-01-24 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Renal Insufficiency, Acute; Cardiac Surgery Associated - Acute Kidney Injury
Keywords: acute kidney injury; early detection; renal artery; doppler ultrasonography; cardiopulmonary bypass
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Patients without CCI-AKI: atients who did not develop CCI-AKI postoperatively (n=64). Observational data collected on demographics, RRI, intraoperative and postoperative factors.
- Group 2: Patients with CCI-AKI: Patients who developed CCI-AKI postoperatively (n=26). Data includes renal failure staging, RRT requirements, complications, and outcomes.

SUMMARY:
The primary aim of our study was to investigate the role of renal doppler ultrasonography (USG) and preoperative/postoperative renal resistive index (RRI) in the early prediction of AKI. Our secondary aim is to evaluate perioperative parameters that may cause AKI, to determine the duration of intensive care unit (ICU)/hospitalization and 30-day mortality.

DETAILED DESCRIPTION:
Our prospective, observational, cross-sectional study included patients with elective cardiac surgery under general anesthesia with prolonged CRP (>70 min) and aortic cross-clamp (ACC) (>60 min), >18 years of age, without preoperative acute/chronic renal failure, and with preoperative/postoperative RRI measurements. Demographic data, comorbidities, medications, preoperative ejection fraction, admission hematocrit (HCT) and baseline serum creatinine (sCr), type of operation, and preoperative RRI were recorded. Intraoperative operation and CPB/ACC duration, blood product transfusion, urine output, amount of bleeding, fluid balance, use of vasopressor/inotropic agents and diuretics, and complications were recorded. RRI was measured by the same radiologist in the first postoperative hour. Urine output and fluid balance, vasopressor/inotropic agent requirement, diuretic use, sKr, HCT level and blood product transfusion were recorded for 3 days postoperatively. According to KDIGO guidelines, patients who did not develop CCI-AKI were divided into 2 groups as Group 1 (n:64) and patients who developed CCI-AKI were divided into Group 2 (n:26). In Group 2, renal failure stage, duration (acute/chronic) and RRT were recorded. ICU and hospital length of stay, postoperative complications and 30-day mortality were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac surgeries under general anesthesia with prolonged CPB (>70 min) and aortic cross clemp (>60 min) time
* >18 years of age, without preoperative acute or chronic renal failure
* with preoperative and postoperative RRI measurements

Exclusion Criteria:

* Patients with known renal insufficiency,
* Patients with acute renal failure in the last 3 months
* Emergency surgeries,
* Patients with arrhythmia end-stage renal disease and renal transplant
* Patients Patients with short duration of CPB (<70 min) and ACK (<60 min)
* Failed Doppler ultrasonography imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing open heart surgery with cardiopulmonary bypass under general anesthesia
Sampling Method: Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Comparison of preoperative, postoperative renal resistive index [median (min-max)] | Cases between September 2022 and January 2024
  The study aims to evaluate preoperative and postoperative renal resistive index (RRI) values between two groups. The renal resistive index (RRI) is a measure of renal vascular resistance obtained via Doppler ultrasound. . RRI values of 0.7 or higher are associated with worse renal outcomes, as they indicate increased vascular resistance. Statistical analyses will be performed to compare preoperative and postoperative RRI values between the groups.
Preoperative-postoperative percentage change of RRI (∆RRI) between two groups | Cases between September 2022 and January 2024
  The study aims to evaluate percentage change RRI (∆RRI) between two groups. Statistical analyses will be performed to compare magnitude of change in ∆RRI, between the groups.
Postoperative RRI ROC analysis | Cases between September 2022 and January 2024
  The study aims to assess the utility of postoperative renal resistive index (RRI) in predicting the development of cardiac surgery-associated acute kidney injury (CSA-AKI). Receiver operating characteristic (ROC) analysis will be employed to determine the discriminatory power of postoperative RRI and identify an optimal cut-off value for predicting CSA-AKI. Sensitivity, specificity, and predictive probabilities associated with the cut-off value will be evaluated.
Postoperative grouping of patients according to KDIGO criteria | Cases between September 2022 and January 2024
  The study plans to include 90 patients, categorized into two groups based on the KDIGO criteria for acute kidney injury (AKI): patients who do not develop cardiac surgery-associated AKI (CSA-AKI) and patients who do develop CSA-AKI. To analyze differences between the groups, specific clinical and biochemical parameters will be assessed and reported as separate outcome measures. These parameters will include [specific measurements, e.g., serum creatinine levels (mg/dL), estimated glomerular filtration rate (eGFR, mL/min/1.73m²), and urine output (mL/kg/hour)]. Each parameter will be assessed using standard laboratory or clinical methods, with units of measurement specified for each outcome. If multiple measurements are aggregated to generate a single outcome (e.g., BMI calculated from weight and height), this will be clearly described in the analysis.

SECONDARY OUTCOMES:
Hematocrit Change over Time [median (min-max)] | Cases between September 2022 and January 2024
  The study will assess changes in intraoperative hematocrit (Hct) values over time. Hct levels will be measured at predefined stages of the operation, including the warm-up period, and comparisons between the groups will be conducted to evaluate potential differences.
Distribution of Intraoperative Urine Output (mL) [median (min-max)] | Cases between September 2022 and January 2024
  The study will evaluate intraoperative urine output (mL) between the groups. Urine output will be measured at three distinct time points: before cardiopulmonary bypass (CPB), during CPB, and after CPB.
Distribution of Intraoperative Administered Fluids (mL) [median (min-max)] | Cases between September 2022 and January 2024
  The study will evaluate the volume of fluids administered intraoperatively in both groups. The total volume of fluids administered (mL) during the intraoperative period will be recorded and analyzed.
Distribution of Intraoperative Fluid Balance (mL) Between Groups [median (min-max)] | Cases between September 2022 and January 2024
  Fluid balance will be assessed intraoperatively as the difference between the total volume of fluids administered and the total output (urine and other losses). This parameter will be reported in mL and analyzed to identify differences between the groups.
Comparison of Urine Output in the First 3 Postoperative Days Between and Within Groups [mean ± SD] | Cases between September 2022 and January 2024
  The study will evaluate postoperative urine output in both groups over the first three days following surgery. Urine output will be measured daily, and comparisons will be conducted to assess differences between the groups at each time point.
Comparison of Fluid Balance in the First 3 Postoperative Days Between and Within Groups[mean ± SD] | Cases between September 2022 and January 2024
  The study will analyze 24-hour fluid balance values for the first three postoperative days. Daily fluid balance values will be compared between the groups to identify potential differences at each time point.
Intergroup and Intragroup Comparison of Postoperative First 3 Days sKr Values [median (min-max)] | Cases between September 2022 and January 2024
  The study will assess serum creatinine (sCr) levels over the first three postoperative days. Comparisons will be made between the groups to evaluate differences in sCr values at each time point.
Comparison of Postoperative Duration of ICU Stay, Duration of Hospitalization Between Groups (day) [median (min-max)] | Cases between September 2022 and January 2024
  This outcome measure will evaluate and compare the postoperative duration of ICU stay and the total duration of hospitalization (in days) between the two groups. The duration of ICU stay will be recorded as the total number of days patients spend in the ICU after surgery, while the duration of hospitalization will include the total number of days from admission to discharge. Both outcomes will be reported as median values (with minimum and maximum ranges) for each group. Statistical analyses will be conducted to identify any significant differences between the groups.
Comparison of duration of postoperative mechanical ventilation (hour) [median (min-max)] | Cases between September 2022 and January 2024
  The study will compare the duration of postoperative mechanical ventilation between the groups. This outcome measure will record the total time (in hours) that patients require mechanical ventilation following surgery. Data will be presented as the median value with a range (minimum to maximum) to account for variability. Statistical analyses will be conducted to identify any significant differences in mechanical ventilation duration between the groups.
Comparison of Postoperative prolonged mechanical ventilation (>6 hours) Between Groups [median (min-max)] | Cases between September 2022 and January 2024
  This outcome measure evaluates the incidence of prolonged postoperative mechanical ventilation, defined as ventilation duration exceeding 6 hours, in each group. The data will be reported as the percentage of patients requiring prolonged mechanical ventilation, along with the median duration of ventilation and its range (min-max). Statistical comparisons will be conducted to determine significant differences between the groups.
Comparison of Postoperative 1-month mortality rate Between Groups [median (min-max)] | Cases between September 2022 and January 2024
  The study will compare the postoperative 1-month mortality rate between the groups. This outcome measure represents the proportion of patients who die within 30 days after surgery. The mortality rate will be reported as a percentage and summarized using median (min-max) values for each group. Statistical analyses will be conducted to evaluate differences in 1-month mortality rates between the groups.
Postoperative Blood and Blood Products Transfusion, n (percent) | Cases between September 2022 and January 2024
  The study will assess the number of erythrocyte suspension (ES) transfusions required in each group. Subgroup analysis will be conducted to evaluate the incidence of transfusion requirements between the groups.
KDIGO Stages in Patients with Renal Failure, n (percent) | Cases between September 2022 and January 2024
  The study will assess the incidence of acute kidney injury (AKI) based on the Kidney Disease: Improving Global Outcomes (KDIGO) classification. The KDIGO staging system categorizes AKI into three stages (Stage 1 to Stage 3) based on serum creatinine levels and urine output. Higher stages indicate worse outcomes, reflecting greater severity of renal dysfunction. The study will also evaluate the occurrence of renal failure, the need for renal replacement therapy (RRT), and the rate of permanent renal failure. The timing of AKI onset and the need for interventions such as continuous renal replacement therapy (CRRT) or hemodialysis during the postoperative period will be monitored.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa High Specialization Training and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bossard G, Bourgoin P, Corbeau JJ, Huntzinger J, Beydon L. Early detection of postoperative acute kidney injury by Doppler renal resistive index in cardiac surgery with cardiopulmonary bypass. Br J Anaesth. 2011 Dec;107(6):891-8. doi: 10.1093/bja/aer289. Epub 2011 Sep 22. PMID 21940396
- [Background] Karim HM, Yunus M, Saikia MK, Kalita JP, Mandal M. Incidence and progression of cardiac surgery-associated acute kidney injury and its relationship with bypass and cross clamp time. Ann Card Anaesth. 2017 Jan-Mar;20(1):22-27. doi: 10.4103/0971-9784.197823. PMID 28074790